CLINICAL TRIAL: NCT00337792
Title: A Randomized Clinical Trial Comparing Oral Conscious Sedation With Intravenous Conscious Sedation for First Trimester Surgical Abortion
Brief Title: Comparing the Effectiveness of Oral Versus Intravenous Pain Medicine for Suction Curettage (D&C)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB review at 50% recruitment, further recruitment unlikely to change result
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Jane Doe, Planned Parenthood League of MA
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-002284/1
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Undesired Pregnancy
MeSH Terms: interventions — Oxycodone; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oxycodone + lorazepam versus fentanyl + midazolam

SUMMARY:
The main objective of this study is to determine the equivalency of oral conscious sedation and intravenous conscious sedation for first trimester surgical abortion. We hypothesize that oral conscious sedation will be equivalent to intravenous conscious sedation for pain control. Additional objectives include describing subject satisfaction with each method of pain control and characteristics of each method such as side effect profile, recovery room time, and postoperative pain.

DETAILED DESCRIPTION:
The main objective of this study is to determine the equivalency of oral conscious sedation (oxycodone 10mg PO plus lorazepam 1mg SL) and intravenous conscious sedation (fentanyl 100 µg plus midazolam 2mg) for first trimester surgical abortion. We hypothesize that oral conscious sedation will be equivalent to intravenous conscious sedation as defined by ± 1 point on a 21-point pain scale. Subsidiary objectives include describing subject satisfaction with each method of pain control and characteristics of each method such as side effect profile, recovery room time, and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Undesired pregnancy between 6 0/7-12 6/7 weeks gestation.
* Has already signed consent for pregnancy termination.
* Eligible for IV sedation per clinic protocol.

Exclusion Criteria:

* Under 120 lbs.
* Allergies to any of the drugs being studied.
* Chronic narcotics, barbiturates or benzodiazepine use within the past year.
* History of IV drug use within the last year.
* Inability to give informed consent.
* Does not speak English or Spanish and does not have translator for all study procedures
* Previously participated in study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain scale

SECONDARY OUTCOMES:
Measures of satisfaction, side effects, recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Jane Doe, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Allen RH, Fitzmaurice G, Lifford KL, Lasic M, Goldberg AB. Oral compared with intravenous sedation for first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):276-83. doi: 10.1097/AOG.0b013e3181938758. PMID 19155895